CLINICAL TRIAL: NCT05695573
Title: Determination of Uromodulin as a Potential Biomarker of Diabetic Kidney Disease
Brief Title: Assessment of Urinary Uromodulin and the Corresponding Gene Expression as a Biomarker of Diabetic Nephropathy
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Collaborators: Ain Shams University (Other)
Responsible Party: Principal Investigator, Shaimaa Ibrahim Barr, Tanta, Egypt, Ain Shams University
Other Study IDs: DN UMOD
Record Dates: First submitted 2023-01-13; First posted 2023-01-25 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Diabetic Nephropathy
MeSH Terms: conditions — Diabetic Nephropathies | interventions — Blood Urea Nitrogen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine samples: first morning samples were collected 3ml for ACR 15ml was stored at -80 ℃ until the time of exosome isolation 6ml of peripheral venous blood were collected 2ml of venous blood was collected in an EDTA vacutainer tube for determination of HbA1c.
  1ml of venous blood was drawn from each subject 2hrs after meal for postprandial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Controlgroup: 25 healthy volunteer as a control
  Interventions: Diagnostic Test: ACR, fasting, postprandial blood glucose ,HbA1c, creatinine, cystatin-C, BUN, Na, K , lipid profile
- diabetic patients with normoalbuminuria: Consisted of 25 type 2 diabetic patients with normoalbuminuria (levels <30 mg/g creatinine)
  Interventions: Diagnostic Test: ACR, fasting, postprandial blood glucose ,HbA1c, creatinine, cystatin-C, BUN, Na, K , lipid profile
- diabetic patients with microalbuminuria: Consisted of 25 type 2 diabetic patients with microalbuminuria (between 30-300 mg/g creatinine).
  Interventions: Diagnostic Test: ACR, fasting, postprandial blood glucose ,HbA1c, creatinine, cystatin-C, BUN, Na, K , lipid profile
- diabetic patients with macrolbuminuria: Consisted of 25 type 2 diabetic patients with macroalbuminuria (levels >300 mg/g creatinine)
  Interventions: Diagnostic Test: ACR, fasting, postprandial blood glucose ,HbA1c, creatinine, cystatin-C, BUN, Na, K , lipid profile

INTERVENTIONS:
Diagnostic Test: ACR, fasting, postprandial blood glucose ,HbA1c, creatinine, cystatin-C, BUN, Na, K , lipid profile — Use the ACR to divide diabetic patients to 3groups not normoalbuminuria, microalbuminuria, macroalbuminuria to evaluate the urinary uromodulin level and its exosomal umod mRNA as a potential biomarker of Diabetic nephropathy diagnosis

SUMMARY:
Detecting diabetes-related kidney diseases early is crucial to prevent end-stage renal disease (ESRD). Existing biomarkers' specificity and sensitivity vary, emphasizing the need for novel markers. This research assesses urinary uromodulin levels and its gene expression, aiming to identify a potential marker for early diabetic nephropathy (DN) detection in type 2 diabetes patients. Uromodulin, encoded by the UMOD gene, is expressed mainly in the thick ascending limb of Henle's loop epithelial cells, making it a promising candidate for early DN detection and progression towards ESRD, potentially reducing chronic kidney disease prevalence.

DETAILED DESCRIPTION:
Introduction:

Diabetes mellitus (DM) is a metabolic disorder characterized by elevated blood glucose levels resulting from deficiencies in insulin secretion, insulin action, or both. Prolonged hyperglycemia associated with diabetes can lead to lasting damage and dysfunction in various organs, including the eyes, kidneys, nerves, heart, and blood vessels (American Diabetes Association, 2008).

Among the complications of diabetes, diabetic nephropathy (DN) stands out as a significant contributor to chronic kidney disease (CKD) (Macisaac et al., 2014). Pathophysiologically, DN progresses from an early phase featuring glomerular hypertrophy, hyperfiltration, and microalbuminuria to an advanced phase marked by progressive glomerulosclerosis, increased urinary albumin excretion (UAE), and impaired renal function (Schrijvers et al., 2004).

Traditionally, DN severity is assessed by measuring urine albumin levels, with persistent microalbuminuria (30-300 mg/24 hr) or macroalbuminuria (>300 mg/24 hr) serving as markers and predictors of DN and its progression to end-stage renal disease (Adler et al., 2003).

Current practices in biomarker use for DN diagnosis show conflicting results regarding sensitivity and specificity in recent studies. Therefore, it is imperative to identify novel biomarkers for early DN detection and progression to reduce the prevalence of chronic kidney diseases in the population (Carole et al., 2017).

Uromodulin, also known as Tamm-Horsfall protein, is an 85 kDa glycoprotein normally secreted by epithelial cells lining the thick ascending limb (TAL) of Henle's loop and early distal tubule. It is released through proteolytic cleavage of glycosylphosphatidylinositol (GPI)-anchored protein, primarily localized to the apical plasma membrane. Uromodulin levels undergo significant changes in urinary excretion during pathological conditions, making it a valuable marker for renal disease

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic patients with not no album in ur is, micoalbuminuria and macroalbuminuria

Exclusion Criteria:prescence of non diabetic or obstructive kidney disease,

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients were selected from those admitted to the Internal Medicine Department and outpatients of Tanta University Hospital
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-07-05 (Actual); Primary Completion 2022-04-28 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Determination the level of urinary uromodulin as a potential biomarker for early prediction of DN | June, 2022
  Evaluate the level of urinary uromodulin in the 3 diabetic group comparing with each other and compare them to the control group and correlate these results with other kidney biomarker
Determine the urinary exosomal UMODmRNA gene expression | June, 2022
  Isolation of urinary exosomes and extraction the UMOD mRNA from these exosoms and determine the fold change of the exosomal UMOD mRNA between the diabetic groups and control group and correlate it with the urinary uromodulin level and other kidney biomarker

CONTACTS AND LOCATIONS:
Overall Officials: Tarek M mohamed, prof, Study Director — Faculty of science, tanta university; Eman M Abd elAzeem, prof, Study Director — faculty of science, Ain shams University
Locations (1):
- Tanta university hospital, faculty of science, tanta university, Tanta, Al Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- See also: Related Info — http://pubmed.ncbi.nlm.nih.gov/29779026/